CLINICAL TRIAL: NCT04726605
Title: Translation and Validation of the Turkish Version of the Postoperative Quality of Recovery Score QoR-15
Brief Title: Turkish Version of the Postoperative QoR-15
Acronym: QoR-15T
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Umut Kara, Consultant, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: 2020/246
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Surgery; Cross-Cultural Comparison; Postoperative Period; Recovery of Function
Keywords: Questionnaire Quality-of-recovery 15 (QoR-15)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patient perceived quality of recovery is an important outcome after surgery and should be measured in clinical trials. The QoR-15 was designed to measure quality of recovery after surgery. It provided an efficient evaluation of the postoperative quality of recovery. The primary objectives of this study is to translate the original QoR-15 questionnaire into Turkish, and do a full psychometric evaluation of the Turkish version. We will test its validity, reliability, responsiveness, and clinical acceptability and feasibility, with patients undergoing abdominal, thoracic, orthopedic, gynecological, urologic, eye and ENT surgery, in the University of Health Sciences, Gülhane Education and Rraining Hospital Ankara, Türkiye.

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 years old
* underwent selective or day surgery with general anesthesia (including all surgical categories except heart and vascular surgery)
* able to complete the QoR-15T in Turkish
* agreed to provide written informed consent to participate

Exclusion Criteria:

* aged < 18 years old
* patients with a neuropsychiatric disturbance
* not agreed to provide written informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted for any type of scheduled surgery with general anesthesia except heart and vascular surgery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery 15 Score | 24 hours after surgery
  Postoperative Quality of Recovery 15 in Turkish scale (QoR-15T)

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Gülhane Education and Training Hospital, Etlik, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Lyckner S, Boregard IL, Zetterlund EL, Chew MS. Validation of the Swedish version of Quality of Recovery score -15: a multicentre, cohort study. Acta Anaesthesiol Scand. 2018 Aug;62(7):893-902. doi: 10.1111/aas.13086. Epub 2018 Feb 7. PMID 29417552